CLINICAL TRIAL: NCT06121661
Title: APPRAISE 2.0: Live Trial of the APPRAISE Trauma Decision Support System
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Andrew Tomas Reisner (Other)
Responsible Party: Sponsor-Investigator, Andrew Tomas Reisner, Principal Investigator; Associate Prof. of Emergency Medicine, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2022P001136
Record Dates: First submitted 2023-10-18; First posted 2023-11-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Wounds and Injuries
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- APPRAISE cases (Experimental): Trauma patients for which APPRAISE system was used
  Interventions: Device: APPRAISE Trauma Clinical Decision Support System

INTERVENTIONS:
Device: APPRAISE Trauma Clinical Decision Support System — Real-time bedside decision-support system for trauma patient management

SUMMARY:
This is a pilot evaluation of the APPRAISE trauma decision-support software system ("the System"). The specific objections are as follows:

1. Evaluate the robustness of the System (i.e., whether the software performs in real-time in accordance with a priori technical specifications during real-time clinical use);
2. Evaluate whether the real-time display of the System causes distraction or confusion to clinicians treating the trauma patient such that its risks exceed its benefits;
3. Collect pilot data to allow for a statistical power analysis to design a future clinical trial evaluating efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 yrs) Emergency Department (ED) patient
* Triaged to the "Acute" area of the ED. (The "Acute" area is the designated area for ED patients with potential or established critical illness. Triage to Acute is a routine ED operation that is performed based on departmental guidelines and the professional judgement of an experienced triage nurse).
* Clinical concern for acute injury (based on either an explicitly chief complaint of acute injury, or clinical team with documented concern for acute injury as a relevant part of patient presentation).

Exclusion Criteria:

* Prisoners
* Patients known to be pregnant, based on patient report, physical exam, or bedside ultrasound
* Patients wearing an "EFIC Opt-Out" bracelet
* Any concern about the suitability of the software system for a specific patient by any clinician involved in the patient's ED care, or by the patient themselves (or by any LAR [lawfully authorized representative] of the patient).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-02-21 (Actual); Primary Completion 2027-12-14 (Estimated); Study Completion 2028-12-14 (Estimated)

PRIMARY OUTCOMES:
Software session with error messages or critical software errors | From patient arrival in the Emergency Department through enrollment, protocol initiation, and protocol completion (which is typically 30 min after protocol initiation).
  Each time the software is used ("session"), a log file is generated. We will quantify how many sessions generate error messages or critical software errors.
Clinician surveys that the software negatively affected patient care | From patient arrival in the Emergency Department through enrollment, protocol initiation, and protocol completion (which is typically 30 min after protocol initiation)
  Each time the software is used, clinicians are surveyed whether the software negatively affected patient care, in their professional judgement
Clinician surveys that the software positively affected patient care | From patient arrival in the Emergency Department through enrollment, protocol initiation, and protocol completion (which is typically 30 min after protocol initiation)
  Each time the software is used, clinicians are surveyed whether the software negatively affected patient care, in their professional judgement
Clinician surveys that ongoing use of the software poses risks that exceeds benefits | From patient arrival in the Emergency Department through enrollment, protocol initiation, and protocol completion (which is typically 30 min after protocol initiation)
  Each time the software is used, clinicians are surveyed whether ongoing use of the software poses risks that exceeds benefits

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Reisner, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States